CLINICAL TRIAL: NCT03097913
Title: Kaohsiung Medical University Chung-Ho Memorial Hospital
Brief Title: Technique Using Trachway to Safely Navigate Endotracheal Tube Through Nasal Cavity
Acronym: video-stylet
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(II)_20160112
Record Dates: First submitted 2017-02-28; First posted 2017-03-31 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2017-03

CONDITIONS: Nasotracheal Intubation
Keywords: nasotracheal intubation; video-stylet; nasal cavity injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- video-stylet tube assembly: patients who undergo oxo-maxillofacial surgery with nasotracheal intubation general anesthesia are recruited
  Interventions: Device: video-stylet

INTERVENTIONS:
Device: video-stylet — recording each video-stylet endotracheal tube assembly advanced through the selected nasal cavity

SUMMARY:
To investigate the double curve endotracheal tube safely navigate through nasal cavity under guidance of a video-stylet.

DETAILED DESCRIPTION:
we enrolled consecutive patients undergoing oxo-maxillofacial surgery by using video-stylet to establish airway and realize the tube angle changes while advancement, however, patients who did not inform or refuse to enroll into the study still use the video-stylet establish airway. the technique to use videostylet-tube assembly to establish airway is a commonly clinical practice in our hospital.

In general, the endotracheal tube goes through nasal cavity blindly either assist with traditional laryngoscope or video-laryngoscope. Tube advances through selected nasal cavity by using a video-stylet is able to prevent from damages of the abnormal turbinates and tissue mucosa. In addition, we are able to record the stylet angle into nostril, shift axis angle in nasal cavity to prevent orifice and side hole from damaging tissues while tube-stylet assembly advancement, and the angle ranges from initiate intubation to tube advanced into trachea.

the selected nostril is determined by Otolaryngologist who is not aware of the study.

ELIGIBILITY:
Inclusion Criteria:

* patients undergo regular operation of oro-maxillofacial surgery

Exclusion Criteria:

* easily nasal bleeding, mouth limited (opening mouth < 3cm), hypertension, diabetes, chronic sinusitis with operative history, patients unwilling to be included.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing regular oro-maxillofacial surgery are included in the study from a medical university hospital (medical center)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
assessment nasal cavity and nasopharyngeal tissues damages | 5-10 minutes
  using video-stylet to safely navigate through selected nasal cavity and advancement into trachea

SECONDARY OUTCOMES:
video-stylet forward trend and angle changes during intubation | 5-10 minutes
  put tube-stylet assembly into selected nostril needs change the vectors while advancement
postoperative nasal damages | 24 hours
  measurement of nasal bleeding and nasal congestion and nasal pain

CONTACTS AND LOCATIONS:
Overall Officials: kuang I Cheng, MD, PhD, Study Director — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Department of Anesthesiology, Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsu HT, Lin CH, Tseng KY, Shen YC, Chen CH, Chuang WM, Cheng KI. Trachway in assistance of nasotracheal intubation with a preformed nasotracheal tube in patients undergoing oral maxillofacial surgery. Br J Anaesth. 2014 Oct;113(4):720-1. doi: 10.1093/bja/aeu334. No abstract available. PMID 25236899
- [Result] Lee MC, Tseng KY, Shen YC, Lin CH, Hsu CW, Hsu HJ, Lu IC, Cheng KI. Nasotracheal intubation in patients with limited mouth opening: a comparison between fibreoptic intubation and the Trachway(R). Anaesthesia. 2016 Jan;71(1):31-8. doi: 10.1111/anae.13232. Epub 2015 Oct 12. PMID 26460721